CLINICAL TRIAL: NCT02047552
Title: A Randomized Controlled Pilot Study of Goal-directed Iron Supplementation of Anemic, Critically Ill Trauma Patients With Functional Iron Deficiency, With and Without Oxandrolone
Brief Title: RCT of Goal-directed Iron Supplementation of Anemic, Critically Ill Trauma Patients, With and Without Oxandrolone
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No Participants enrolled
Sponsor: Denver Health and Hospital Authority (Other)
Responsible Party: Principal Investigator, Fredric Pieracci, Assistant Professor of Surgery, Denver Health and Hospital Authority
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14-0167
Record Dates: First submitted 2014-01-26; First posted 2014-01-28 (Estimated); Last update posted 2019-04-03 (Actual); Status verified 2019-04

CONDITIONS: Functional Iron Deficiency; Trauma; Anemia
Keywords: trauma; iron; anemia; red blood cell transfusion
MeSH Terms: conditions — Wounds and Injuries; Anemia | interventions — Ferric Oxide, Saccharated; Oxandrolone; Steroids

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Iron sucrose (Active Comparator): Iron sucrose 100 mg IV will be dosed daily for up to seven days if, on morning laboratory analysis, (1) TSAT < 25%, (2) Serum iron concentration < 150 ug/mL, and (3) Serum ferritin concentration < 1,500 ng/mL. Thus, the maximum possible cumulative dose of iron sucrose over the one-week dosing period will be 700 mg.
  Interventions: Drug: Iron sucrose; Drug: Oxandrolone placebo
- Oxandrolone (Active Comparator): Oxandrolone 10 mg PO q12 hours will be dosed for seven days.
  Interventions: Drug: Oxandrolone; Drug: IV iron placebo
- Iron sucrose + oxandrolone (Experimental): Combination goal-directed iron sucrose (as described in the iron sucrose only arm) and oxandrolone (as described in the oxandrolone only arm) for seven days.
  Interventions: Drug: Iron sucrose; Drug: Oxandrolone
- IV iron placebo and Oxandrolone placebo (Placebo Comparator): 100 mL normal saline in place of iron and similar color and size sugar pill for Oxandrolone placebo
  Interventions: Drug: IV iron placebo; Drug: Oxandrolone placebo

INTERVENTIONS:
Drug: Iron sucrose — Iron sucrose 100 mg IV will be dosed daily for up to seven days if, on morning laboratory analysis, (1) TSAT < 25%, (2) Serum iron concentration < 150 ug/mL, and (3) Serum ferritin concentration < 1,500 ng/mL. Thus, the maximum possible cumulative dose of iron sucrose over the one-week dosing period will be 700 mg.
  Other Names: Fe
  Arms: Iron sucrose; Iron sucrose + oxandrolone
Drug: Oxandrolone — 10 mg PO Q12 hours for seven days
  Other Names: Steroid
  Arms: Iron sucrose + oxandrolone; Oxandrolone
Drug: IV iron placebo — 100 mL normal saline
  Other Names: Fe placebo
  Arms: IV iron placebo and Oxandrolone placebo; Oxandrolone
Drug: Oxandrolone placebo — similar color and size sugar pill
  Other Names: Steroid placebo
  Arms: IV iron placebo and Oxandrolone placebo; Iron sucrose

SUMMARY:
The purpose of this trial is to determine if the combination of goal directed iron supplementation and hepcidin mitigation can safely eliminate both the serum and bone marrow iron debt of anemic, critically ill trauma patients with functional iron deficiency.

DETAILED DESCRIPTION:
The inflammatory response associated with traumatic critical illness rapidly induces a functional iron deficiency, characterized by hypoferremia, decreased transferrin saturation (TSAT), hyperferritinemia, and iron-deficient erythropoiesis (IDE). These derangements in iron metabolism are primarily related to upregulation of the iron regulatory protein hepcidin, which inhibits ferroportin-mediated release of iron from both duodenal enterocytes and macrophages. The resultant functional iron deficiency both contributes to intensive care unit (ICU) anemia and increases the packed red blood cell (pRBCs) transfusion requirement.

Treatment strategies for functional iron deficiency in critically ill patients may be divided broadly into (1) iron supplementation and (2) mitigation of the effects of hepcidin. The goals of treatment are to reverse the serum iron debt, eliminate IDE, improve anemia, and ultimately decrease pRBCs transfusions. Given that approximately 90% of critically ill trauma patients with an ICU length of stay (LOS) ≥ 7 days receive at least one pRBCs transfusion, any strategy that has even a modest impact upon the transfusion requirement is likely to improve overall health outcomes substantially.

Issues surrounding iron supplementation of critically ill patients include formulation, dose, route of administration, hepcidin antagonism, and mitigation of the complications of iron overload, particularly infection. Our first RCT of iron supplementation of critically ill surgical patients compared enteral ferrous sulfate 325 mg thrice daily to placebo (NCT00450177). Although a significant reduction in pRBCs transfusion requirement for the iron group was observed, low injury severity, intolerance of enteral medications, and a predominance of traumatic brain injury limited generalizability. In a second multicenter RCT, we compared intravenous iron sucrose 100 mg thrice weekly to placebo among critically ill trauma patients (NCT01180894, NTI-ICU-008-01) [8]. Iron supplementation using this generic dosing scheme did not impact the serum iron concentration, TSAT, IDE, anemia, or pRBCs transfusion requirement. Rather, iron supplementation accumulated as ferritin as evidenced by a significantly increased serum ferritin concentration in the iron as compared to the placebo group at all time points. Iron supplementation did not increase the risk of infection in either trial, despite a relatively high incidence of marked hyperferritinemia (serum ferritin concentration > 1,000 ng/mL) in the iron group.

The results of these trials suggest that iron supplementation alone, and using a generic dosing scheme, is ineffective. The current pilot trial aims to build upon the findings of the prior two RCTs by incorporating both goal-directed iron supplementation and hepcidin antagonism. The hypothesis is that the combination of goal directed iron supplementation and hepcidin mitigation will safely eliminate both the serum and bone marrow iron debt of anemic, critically ill trauma patients with functional iron deficiency.

ELIGIBILITY:
Inclusion Criteria:

1. Informed consent from patient or patient representative.
2. Trauma patient
3. Anemia (hemoglobin < 12 g/dL).
4. Functional iron deficiency:

   1. Serum iron concentration < 40 ug/dL
   2. TSAT < 25%
   3. Serum ferritin concentration > 28 ng/mL
5. < 72 hours from ICU admission.
6. Expected ICU length of stay ≥ 7 days.

Exclusion Criteria:

1. Age < 18 years.
2. Active bleeding requiring pRBCs transfusion.
3. Iron overload (serum ferritin concentration ≥ 1,500 ng/mL). The serum ferritin concentration is an acute phase reactant that is increased during critical illness regardless of total body iron. Substantial levels of hyperferritinemia (serum ferritin concentration > 1,000 ng/dL) were observed in both NCT00450177 and NCT01180894 without increased risk of infection and despite both low TSAT and IDE. For these reasons, we believe that relative hyperferritinemia (serum ferritin concentration 500 - 1,500 ng/dL) is neither harmful nor indicative of bone marrow iron availability.
4. Infection, defined using US Centers for Disease Control and Prevention (CDC) guidelines, with the exception of ventilator-associated pneumonia (VAP), which is defined as clinical suspicion for pneumonia along with a lower respiratory tract culture with ≥ 105 colony forming units per mL.
5. Chronic inflammatory conditions (e.g., systemic lupus erythematosis, rheumatoid arthritis, ankylosing spondylitis).
6. Pre-existing hematologic disorders (e.g., thalassemia, sickle cell disease, hemophilia, von Willibrand's disease, or myeloproliferative disease).
7. Pre-existing hepatic dysfunction (cirrhosis, non-alcoholic steatohepatitis, hepatitis)
8. Current or recent (within 30 days) use of immunosuppressive agents.
9. Use of any recombinant human erythropoietin formulation within the previous 30 days.
10. Known or suspected carcinoma of the breast or prostate.
11. Nephrosis, the nephrotic phase of nephritis.
12. Hypercalcemia (serum calcium concentration > 10.5 mg/dL).
13. Pregnancy or lactation.
14. Legal arrest or incarceration.
15. Prohibition of pRBCs transfusion.
16. Stay of ≥ 48 hours duration in the ICU of a transferring hospital.
17. History of intolerance or hypersensitivity to either iron or oxandrolone.
18. Moribund state in which death was imminent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Serum iron debt (as measured by the transferrin saturation) | One week
  The transferrin saturation will be measured at baseline and daily thereafter for one week

SECONDARY OUTCOMES:
Bone marrow iron debt (as measured by the zinc protoporphyrin) | one week
  Zinc protoporphyrin will be measured at baseline and daily thereafter for one week
Serum ferritin concentration | one week
  The serum ferritin concentration will be measured at baseline and daily thereafter for one week
serum hepcidin concentration | one week
  The serum hepcidin concentration will be measured at baseline and daily thereafter for one week.
Liver function tests | one week
  Liver function tests will be measured at baseline and daily thereafter for one week.
Erythropoeitin concentration | one week
  The serum erythropoeitin concentration will be measured at baseline and daily thereafter for one week.
Red blood cell transfusion requirement | 28 days
  The incidence and number of red blood cell transfusions will be collected for 28 days.
Hemoglobin | 28 days
  The hemoglobin concentration will be measured at baseline and daily thereafter for 28 days.
Infections | 28 days
  The incidence, types, and number of infections will be collected for 28 days.
All cause mortality | 28 days
  All cause mortality will be collected for 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Fredric M Pieracci, MD, MPH, Principal Investigator — Denver Health Medical Center
Locations (1):
- Denver Health Medical Center, Denver, Colorado, United States